CLINICAL TRIAL: NCT07125118
Title: Self-help Interventions for Parenting Couples Experiencing Couple Distress: Study Protocol for a Randomized Controlled Trial
Brief Title: Self-helpinterventions for Parenting Couples With Couple Distress.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Tea Trillingsgaard, Associate Professor, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSS-2024-018-S2; 157457 (Other Grant/Funding Number: Trygfonden)
Record Dates: First submitted 2025-07-12; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Marital Conflict
Keywords: Self-help intervention; OurRelationship program; internet intervention; bibliotherapy; relationship distress; relationship satisfaction; communication conflict; randomized controlled trial; parents; digital mental health; Vores Parforhold; Couple Distress
MeSH Terms: interventions — Bibliotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The OurRelationship Program (Experimental): Participants assigned to this arm complete a guided self-help program for couples that includes online learning modules, structured couple conversations, and support from a trained coach through five scheduled calls.
  Interventions: Behavioral: The OurRelationship Program
- Bibliotherapy (Experimental): Participants assigned to this arm complete an unguided self-help program for couples using the book "Take Care of Your Relationship" [Pas på Parforholdet] and a reading guide, with planned couple conversations.
  Interventions: Behavioral: Bibliotherapy
- Waitlist (No Intervention): Participants receive no intervention during the study period and are offered access to the OurRelationship Program or Bibliotherapy after the follow-up assessment.

INTERVENTIONS:
Behavioral: The OurRelationship Program — A guided self-help program for couples delivered online over 10 weeks. Participants complete structured learning modules and engage in planned couple conversations focused on improving communication, problem-solving, and emotional connection. Each couple receives support from a trained coach through five scheduled telephone or video calls. The program is designed to be flexible and completed at the couple's own pace within the 10-week period.
  Arms: The OurRelationship Program
Behavioral: Bibliotherapy — An unguided self-help program for couples using the Danish book "Take Care of Your Relationship" [Pas på Parforholdet] and an accompanying reading guide. Couples are encouraged to read assigned sections, engage in planned couple conversations, and apply strategies for improving relationship functioning. The intervention is self-paced and completed over 10 weeks without guidance from a coach or therapist.
  Arms: Bibliotherapy

SUMMARY:
Children whose parents experience high levels of couple distress are at greater risk for emotional, behavioral, and academic problems. This study tests two types of self-help for parenting couples: the OurRelationship program (OR), an online guided program, and couple-focused bibliotherapy (BT), a book-based self-help approach. The investigators will compare these interventions with a waitlist (WL) control group to see which is most effective at reducing communication conflict between partners. They will also examine whether the interventions improve child well-being when problems are present at the start of the study.

A total of 350 parenting couples in Denmark will take part. Eligible couples have at least one child under 18 living at home and report high levels of conflict or relationship distress. Couples will be randomly assigned to OR, BT, or WL. Questionnaires will be completed online before the program, after the program (10 weeks later), and at 3- and 12-month follow-ups.

DETAILED DESCRIPTION:
Children exposed to high levels of couple distress are at increased risk for a range of adjustment problems, including behavioral, emotional, and academic difficulties. These relational burdens can also interfere with adult mental health, the coparenting relationship, and the capacity to provide warm and consistent caregiving. Despite these challenges, many couples delay seeking help until their relationship has seriously deteriorated.

This randomized controlled trial investigates the efficacy of two flexible self-help interventions: the OurRelationship program (OR) and couple-focused bibliotherapy (BT). The investigators hypothesize that OR will outperform BT, which in turn will outperform a waitlist (WL) control in reducing communication conflict-the primary outcome-between baseline and post-intervention. The investigators further hypothesize that any couple intervention (OR or BT) will outperform WL in reducing the impact on child well-being-the secondary outcome-between baseline and post-intervention for children showing such impact at baseline.

Parenting couples (N = 350) with one or more children living at home, who report either high levels of parental conflict or relationship distress, are recruited via municipal family services in 11 or more Danish sites. Participants enroll through an online platform, complete a screener, provide informed consent, and fill out a baseline survey before randomization. Families are randomly assigned in a 1:1:1 ratio to OR, BT, or WL. Online questionnaires are completed at baseline (T1, before randomization), post-intervention (T2, 10 weeks after randomization), and at 3-month and 12-month follow-ups (T3 and T4, respectively).

Dyadic multilevel models, with repeated measures (Level 1) nested within couples (Level 2), will be used to examine group differences in change trajectories across time for continuous outcomes. Including both a BT condition and a WL control allows the investigators to test whether OR offers added benefit over an accessible low-tech self-help option. Apart from the previous pilot, this is the first trial to evaluate OR independently of its developers and the first study conducted outside the United States.

ELIGIBILITY:
Inclusion Criteria:

* Meet at least one of the two following criteria: (1) Destructive conflict: one or both partners report being a victim or perpetrator of at least one act of physical or psychological aggression in the past three months (see exclusion criteria for intimate partner violence) OR (2) Couple distress: One partner scores ≤11 (1 SD below the Danish population mean), or both partners score ≤13 (0.5 SD below the Danish population mean) on the Couple Satisfaction Index-4 (CSI-4).
* Both partners are at least 18 years old.
* Cohabiting.
* Have at least one child under 18 living at home.
* Reside in a participating Danish municipality.
* Completed the baseline survey.
* Able to read and understand Danish.
* Have internet access and a compatible device (computer, tablet, or smartphone).
* Agree not to engage in couple therapy prior to the 3-month follow-up.

Exclusion Criteria:

* Current plans to divorce or separate.
* Ongoing affair.
* Moderate to severe suicidal ideation.
* Recent incident of intimate partner violence resulting in physical injury or fear for the safety or well-being of oneself or one's children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2027-10-09 (Estimated)

PRIMARY OUTCOMES:
Communication Conflict Scale | Pre-assessment (T1) to Post Intervention at Week 10 (T2)
  A 7-item self-report measure assessing how couples handle conflict (e.g., "Small issues suddenly became big arguments"), scored from 1 (Often) to 4 (Never), with higher scores indicating better conflict management. Developed for the Administration for Children and Families Supporting Healthy Marriage Initiative

SECONDARY OUTCOMES:
The Strengths and Difficulties Questionnaire (SDQ) - impact score | Baseline (T1) to Post-intervention at Week 10 (T2)
  The 4-item section of the parent-reported SDQ in which the parent assesses the extent to which a child's difficulties cause distress and interfere with everyday life, scored from 0 (Not at all) to 2 (A lot), with higher scores indicating worse impact.

OTHER OUTCOMES:
Couple Satisfaction Index-4 | Baseline (T1) to Post-intervention at Week 10 (T2)
  A 4-item self-report measure of overall relationship satisfaction, scored from 0 (Not at all / Not at all true) to 5 (Completely / Completely true), with higher scores indicating greater satisfaction.
Responsive Attention Scale | Baseline (T1) to Post-intervention at Week 10 (T2)
  A 10-item self-report measure of perceived partner responsiveness, scored from 1 (Very rarely) to 5 (Very often), with higher scores indicating greater responsiveness.
Intimate Safety Questionnaire | Baseline (T1) to Post-intervention at Week 10 (T2)
  A 4-item self-report measure of perceived safety and comfort with one's partner, scored from 0 (Never) to 4 (Always), with higher scores indicating greater intimacy.
Major Depression Inventory | Baseline (T1) to Post-intervention at Week 10 (T2)
  A 10-item self-report measure of depressive symptoms, scored from 0 (None of the time) to 5 (Always), with higher scores indicating worse symptoms.
Suicidal Behaviors Questionnaire-Revised | Baseline (T1) to Post-intervention at Week 10 (T2)
  A 4-item self-report measure of suicidal ideation and behaviors, with item scores ranging from 1 to 7; higher total scores indicate greater suicide risk.
Family Maltreatment Measure - Partner Violence | Baseline (T1) to Post-intervention at Week 10 (T2)
  A multi-item self-report measure of physical and psychological intimate partner violence, scored from 0 (Never) to 6 (More than 10 times), plus harm/consequence ratings; higher scores indicate greater violence.
WHOQOL-BREF Single Items - Quality of Life, Health, Work Functioning | Baseline (T1) to Post-intervention at Week 10 (T2)
  Three single items from the WHOQOL-BREF assessing satisfaction with quality of life, health, and ability to function at work/home, scored from 1 (Very dissatisfied) to 5 (Very satisfied), with higher scores indicating better quality of life/health/functioning.
Perceived Parenting Capacity | Baseline (T1) to Post-intervention at Week 10 (T2)
  A single item adapted from the WHOQOL-BREF assessing satisfaction with ability to meet children's physical and emotional needs, scored from 1 (Very dissatisfied) to 5 (Very satisfied), with higher scores indicating greater perceived capacity.
Strengths and Difficulties Questionnaire - Internalizing and Externalizing Subscales | Baseline (T1) to Post-intervention at Week 10 (T2)
  Two 5-item parent-report subscales assessing child emotional/internalizing and behavioral/externalizing difficulties, scored from 0 (Not true) to 2 (Certainly true), with higher scores indicating worse symptoms.
Child Sleep Quality Item | Baseline (T1) to Post-intervention at Week 10 (T2)
  A single item assessing whether the child sleeps too little or poorly, scored from 0 (Not true) to 2 (Certainly true), with higher scores indicating poorer sleep quality.
Self-Stigma Item | Baseline (T1) to Post-intervention at Week 10 (T2)
  A single item assessing feelings of inadequacy if unable to solve relationship problems without help, scored from 1 (Strongly disagree) to 5 (Strongly agree), with higher scores indicating greater self-stigma.
Internal and Partner Shame Scales | Baseline (T1) to Post-intervention at Week 10 (T2)
  Two 4-item subscales assessing internal shame and partner-related shame, scored from 0 (Never) to 4 (Always), with higher scores indicating greater shame.

CONTACTS AND LOCATIONS:
Overall Officials: Tea Trillingsgaard, Ph.D, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No
The datasets collected for this study are not publicly available due to institutional restrictions at Aarhus University. However, data may be accessed through collaboration with the principal investigator, provided that the researcher is affiliated with a Danish research institution. All analytic scripts and code used in the study will be made available by the authors upon request to facilitate replication.

REFERENCES:
- [Derived] Trillingsgaard T, Lassen NF, Baucom KJW, Svare LT, Hansen FG, Fentz HN. Self-help interventions for parenting couples experiencing conflict or relationship distress: study protocol for a randomized controlled trial. Trials. 2026 Jan 13. doi: 10.1186/s13063-026-09428-6. Online ahead of print. PMID 41530873
- See also: Official Aarhus University webpage describing the research project, including background, aims, and updates. — https://psy.au.dk/forskning/forskningsprojekter/vores-parforhold
- See also: Public-facing website for the Vores Parforhold initiative, including participant enrollment for the study and access to the self-help programs. — https://voresparforhold.dk